CLINICAL TRIAL: NCT04914429
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Guselkumab (TREMFYA) in Chinese Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of Guselkumab (TREMFYA) in Chinese Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109025; CNTO1959PSO4009 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-06-03; First posted 2021-06-04 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab 100 milligrams (mg) by subcutaneous (SC) injection at Weeks 0, 4, and then every 8 weeks (q8w) through Week 44. Participants will receive matching placebo at Week 16.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo SC injection for guselkumab at Weeks 0, 4, and 12, and then cross over at Week 16 to receive guselkumab 100 mg SC injection at Weeks 16 and 20 and q8w thereafter through Week 44.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab 100 mg will be administered as a SC injection.
  Other Names: TREMFYA
Drug: Placebo — Matching placebo will be administered as a SC injection.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of guselkumab in the treatment of Chinese participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of plaque psoriasis with or without psoriatic arthritis for at least 6 months before screening
* A woman of childbearing potential must have a negative urine pregnancy test at screening and at baseline
* Agree not to receive a live virus or live bacterial vaccination during the study, or within 3 months after the last administration of study drug
* Agree to avoid prolonged sun exposure and avoid use of tanning booths or other ultraviolet (UV) light sources during study
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Has a nonplaque form of psoriasis (example, erythrodermic, guttate, or pustular)
* Has a history of or current signs or symptoms of liver or renal insufficiency (estimated creatinine clearance below 60 milliliter/minute [mL/min]); significant, progressive, or uncontrolled cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Currently has a or has a history of malignancy within 5 year before screening (exceptions are nonmelanoma skin cancer that has been adequately treated with no evidence of recurrence for at least 3 months before the first study drug administration and cervical carcinoma in situ that has been treated with no evidence of recurrence for at least 3 months before screening, or malignancy, which is considered cured with minimal risk of recurrence)
* History of, or ongoing, chronic or recurrent infectious disease, including but not limited to, recurrent sinopulmonary infections, bronchiectasis, recurrent renal/urinary tract infection (example, recurrent pyelonephritis, recurrent cystitis), fungal infection (mucocutaneous candidiasis), an open, draining, or infected skin wound, or an ulcer
* Has previously received guselkumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve a Psoriasis Area and Severity Index (PASI) 90 Response at Week 16 | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response is defined as greater than or equal to (>=)90 percent (%) improvement in PASI score.
Percentage of Participants who Achieve an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16 | Week 16
  The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Number of Participants with Adverse Events (AEs) | Up to Week 56
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Serious Adverse Events (SAEs) | Up to Week 56
  SAE is any untoward medical occurrence that at any dose may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Number of Participants with Reasonably Related Adverse Events (AEs) | Up to Week 56
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs Leading to Discontinuation of Study Intervention | Up to Week 56
  Number of participants with AEs leading to discontinuation of study intervention will be reported.
Number of Participants with Infections | Up to Week 56
  Number of participants with infections including serious infections, and infections requiring oral or parenteral antimicrobial treatment will be reported.
Number of Participants with Serious Hypersensitivity Reactions | Up to Week 56
  Number of participants with serious hypersensitivity reactions (such as anaphylaxis, urticaria, pruritis, angioedema, wheezing, dyspnea, or hypotension) will be reported.
Number of Participants with Injection-site Reactions | Up to Week 56
  An injection-site reaction is any unfavorable or unintended sign that occurs at the study drug injection site. Injection sites will be evaluated for reactions and any injection-site reaction will be recorded as an AE.
Number of Participants with Change from Baseline in Laboratory Abnormalities | Up to Week 56
  Number of participants with change from baseline in laboratory abnormalities (chemistry, hematology) will be reported.
Number of Participants with Laboratory Abnormalities with Maximum Toxicity Grades | Up to Week 56
  Number of participants with laboratory abnormalities (hematology, chemistry) with maximum toxicity grades will be reported. A higher grade indicates more severity.
Number of Participants with Change from Baseline in Vital Signs | Up to Week 56
  Number of participants with change from baseline in vital signs (temperature, heart rate, respiratory rate, blood pressure) will be reported.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve a PASI 100, PASI 75, and PASI 50 Response Over Time | Week 0, 4, 12, 16, 20, 28, 36, 44, 48
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100, 75, and 50 response is defined as 100%, >=75%, and >=50% improvement in PASI score respectively.
Percentage of Participants who Achieve a PASI 90 Response Over Time | Week 0, 4, 12, 16, 20, 28, 36, 44, 48
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response is defined as >=90% improvement in PASI score.
Percentage of Participants who Achieve an IGA Score of Cleared (0) or Minimal (1) Over Time | Week 0, 4, 12, 16, 20, 28, 36, 44, 48
  Percentage of participants who achieve an IGA score of cleared (0) or minimal (1) over time will be reported.
Change from Baseline in Dermatology Life Quality Index (DLQI) Score Over Time | Baseline, Week 4, 16, 28, 48
  The DLQI is a dermatology-specific quality of life (QoL) instrument designed to assess the impact of the disease on a participant's QoL. It is a 10 item patient-reported outcome(s) (PRO) questionnaire that, in addition to evaluating overall QoL, can be used to assess 6 different aspects that may affect QoL: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. The DLQI produces a numeric score that can range from 0 to 30. A higher score indicates more severe disease.
Percentage of Participants who Maintain PASI 90 Response at Week 48 Among Participants who were PASI 90 Responders at Week 16 in Guselkumab Group | Week 48
  The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response is defined as >=90% improvement in PASI score.
Percentage of Participants who Maintain IGA Score of Cleared (0) or Minimal (1) at Week 48 Among Participants who Achieved IGA 0/1 at Week 16 in Guselkumab Group | Week 48
  Percentage of participants who maintain IGA score of cleared (0) or minimal (1) at Week 48 among participants who achieved IGA 0/1 at Week 16 in guselkumab group will be reported.
Percentage of Participants who Achieve an IGA Score of Cleared (0) and an IGA Score of Mild or Better (Less Than or Equal to [<=] 2) Over Time | Week 0, 4, 12, 16, 20, 28, 36, 44, 48
  Percentage of participants who achieve an IGA score of cleared (0) and an IGA score of mild or better (<=2) over time will be reported.
Percentage of Participants who Achieve a DLQI Score of 0 or 1 Over Time Among Participants with Baseline DLQI Greater Than (>) 1 | Week 0, 4, 16, 28, 48
  Percentage of participants who achieve a DLQI score of 0 or 1 over time among participants with baseline DLQI >1 will be reported.
Percentage of Participants With a Reduction of 5 or More Points in DLQI Score Over Time | Week 0, 4, 16, 28, 48
  Percentage of participants with a reduction of 5 or more points in DLQI score over time will be reported.
Percent Change from Baseline in Nail Psoriasis Severity Index (NAPSI) Over Time Among Participants with Nail Psoriasis at Baseline | Baseline, Week 16, 28, 36, 48
  The NAPSI is an index used for assessing and grading the severity of nail psoriasis. A target nail representing the worst nail psoriasis is divided into quadrants and is graded for nail matrix psoriasis (pitting, leukonychia, red spots in the lunula, and nail plate crumbling) and nail bed psoriasis (onycholysis, splinter hemorrhages, oil drop discoloration, and nail bed hyperkeratosis), each on a scale of 0-4 (A higher score indicates more severity). The sum of these scores is the total NAPSI score (0=no psoriasis to 8=psoriasis present in all 4 quadrants of the target nail).
Percentage of Participants with an Scalp-Specific Investigator Global Assessment (ss-IGA) Score of Absence of Disease (0) or Very Mild Disease (1) Over Time Among Participants with Scalp Psoriasis and an ss-IGA Score >=2 at Baseline | Week 0, 16, 28, 36, 48
  The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. The lesions are assessed in terms of the clinical signs of redness, thickness, and scaliness which are scored as: absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), and severe disease (4).
Serum Concentration of Guselkumab Over Time | Week 0, 4, 16, 20, 36, 44, 56
  Serum concentrations of guselkumab over time will be reported.
Number of Participants with Antibodies to Guselkumab | Week 0, 16, 44, 56
  Number of participants with antibodies to guselkumab through week 56 will be reported.
Maximum Titer of Antibodies to Guselkumab Through Week 56 | Week 0, 16, 44, 56
  Maximum titer of antibodies to guselkumab through Week 56 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- China (26):
  - Peking University Third Hospital, Beijing
  - Beijing Tongren Hospital, CMU, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The second Xiangya Hospital of Central South University, Changsha
  - West China Hospital,Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing
  - Fujian Medical University, Fuzhou
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou
  - The 1st affiliated hospital of Anhui Medical University, Hefei
  - Skin Disease Hospital of Shandong Province, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Hospital of Dermatology, Chinese Academy of Medical Science, Nanjing
  - Shanghai Ruijin Hospital, Shanghai
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai skin disease hospital, Shanghai
  - University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan province people's hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Huang K, Geng S, Tao X, Sun L, Ji C, Yang B, Lu Y, Xiao R, Zhang C, Zhang F, Lu Q, Zheng J, Wang H, Shi Y, Li Z, Yan W, Zhang L, Tao J, Zhang S, Yang X, Cheng H, Xu J, Su J, Zhang Z, Song Z, Wang L, Wang R, Zhang T, Zhao W, Huang Y, Chen M, Dong Z, Lyu S, Zheng M. Efficacy and safety of guselkumab in Chinese patients with moderate-to-severe plaque psoriasis: A randomized, double-blind, placebo-controlled trial. Chin Med J (Engl). 2025 Sep 8. doi: 10.1097/CM9.0000000000003771. Online ahead of print. PMID 40921728